CLINICAL TRIAL: NCT02812316
Title: Study to Evaluate the Safety and Efficacy of HI-BRITE Large Diameter Rigid Gas Permeable Contact Lens (Hexafocon b) Test When Worn on a Daily Wear Basis in the Correction of Myopia/Hyperopia/Astigmatism/Presbyopia/ and Irregular Cornea.
Brief Title: Study to Evaluate the Safety and Efficacy of HI-BRITE Large Diameter Rigid Gas Permeable Contact Lens
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Taipei Medical University Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 201210038
Record Dates: First submitted 2016-02-26; First posted 2016-06-24 (Estimated); Last update posted 2017-04-27 (Actual); Status verified 2016-11

CONDITIONS: Refractive Errors
Keywords: Myopia; Scleral lens; Astigmatism; Presbyopia
MeSH Terms: conditions — Refractive Errors; Myopia; Astigmatism; Presbyopia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Scleral lenses (Experimental): Subjects who meet all eligible requirements for entry into the study will be instructed to insert the Hi-Brite Large Diameter Rigid Gas Permeable contact lens in daily wear basis for clinical evaluation purposes.
  Interventions: Device: HI-BRITE Large Diameter Rigid Gas Permeable Contact Lens

INTERVENTIONS:
Device: HI-BRITE Large Diameter Rigid Gas Permeable Contact Lens — Approximately At least one hundred and forty (140) subjects (280 eyes) will be enrolled in this study at approximately two (2) clinical sites in Taiwan. All subjects will be fitted for and dispensed study lenses by each Investigator.

SUMMARY:
Study to evaluate the safety and efficacy of HI-BRITE large diameter rigid gas permeable contact lens (hexafocon b) test when worn on a daily wear basis in the correction of myopia/hyperopia/astigmatism/presbyopia/ and irregular cornea.

DETAILED DESCRIPTION:
Subjects who meet all eligible requirements for entry into the study will be instructed to insert the Hi-Brite Large Diameter Rigid Gas Permeable contact lens in daily wear basis for clinical evaluation purposes.

Treatment period: 6 months

ELIGIBILITY:
Inclusion criteria:

* Ametropic or irregular cornea subjects who need to wear spectacle lens or contact lens in their daily life.
* Is of age at least 20 years old and no older than 65 years old capacity to volunteer.
* Has read and signed the Informed Consent Form or waiver. (4) Has myopia or hyperopia -20.00D～+20.00D, astigmatism -0.25~-4.00D, or presbyopia +1.00D～+3.50D.
* Irregular cornea subjects include keratoconus, high astigmatism (>-4.00D) or post-refractive surgery patients.
* No active ocular disease, infection or any disorder of eyelids and conjunctiva.
* Has reasonable expectation of improvement in visual acuity with the test lenses.
* Is willing and able to follow subject instructions and meet the protocol -specified visit schedule. (If subjects missed any visit, they must be discontinued from the study.) (9) Agrees to wear the test lenses at a daily wear basis. (10) Willing to adapt wearing GP contact lens.

Exclusion criteria:

The subject is ineligible for entry into the study if the subject

* Has any systemic disease affecting ocular health.
* Is using any systemic or topical medications that will, in the Investigator's opinion. Affect ocular physiology or lens performance within one (1) week before entering this study.
* Has an active ocular disease or has ever used systemic steroid or any other medicine that may affect significant on vision or healing.
* Has any Grade 2 or greater finding listed in the Quantification of Slit Lamp Observations Form. Subjects with corneal infiltrates, however, of ANY GRADE, are not eligible.
* Has any "Present" finding listed in the Quantification of Slit Lamp Observations that, in the Investigators' judgment, interferes with contact lens wear.
* Has any scar or neovascularization within the central 4mm of the cornea. Subjects with minor peripheral corneal scarring that, in the Investigator's judgment, does not interfere with contact lens wear are eligible for this study.
* Severe dry eye (Schirmer Test<5mm/5min)
* Corneal keratitis
* Is aphakic
* Had undertaken the following surgery: Retina, Glaucoma, Cataract surgery.
* Is amblyopic, BSCVA can't achieve (include) 20/40(0.5) when wear trial lenses.
* Allergy to contact lens solution.
* ls participating in any other clinical research study.
* Pregnancy or Breast-feeding.

Ages: 20 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 136 (Actual)
Dates: Start 2014-08; Primary Completion 2017-02 (Actual); Study Completion 2017-10 (Estimated)

PRIMARY OUTCOMES:
The success rate of the vision with correction | Wearing the contact lens for 6 months
  * Ametropic group: Subjects wear their lens for at least 6 hours/day and 5 days/ week after visit 9, Distance Lens VA is not less than 20/25 and 90% subjects' VA decreased less than 2 lines with Snellen's chart at the last visit.
  * Irregular Cornea Group: Subjects wear their lens for at least 6 hours/day and 5 days/ week after visit 9, Distance Lens VA is not less than 20/40 and 80% subjects' VA decreased less than 2 lines with Snellen's chart at the last visit.

SECONDARY OUTCOMES:
The effectiveness of each visit | wearing the contact lens for 6 months
  * Ametropic group: To assess each subject for the lens satisfied / problem and assess each time of the vision with correction; the ratio of ametropic correcting vision of 20/25 subjects.
  * Irregular Cornea Group: To assess each subject for the lens satisfied / problem and assess each time of the vision with correction; the ratio of the irregular cornea corrected visual acuity of 20/40 subjects.
The rate of Treatment-Emergent Adverse Events to assess the safety of each visit | wearing the contact lens for 6 months
  To assess the rate of adverse reactions, the proportion of corneal ulcers, the proportion of continuous stroma edema, significant proportion of corneal staining of luciferase, the proportion of corneal infections, the proportion of persistent inflammation of the eyelids, and the proportion of other eye discomfort.

CONTACTS AND LOCATIONS:
Overall Officials: Tsung-Jen Wang, Dr., Principal Investigator — Taipei Medical University Hospital
Locations (1):
- Taipei Medical University Hospital, Taipei, Taiwan

IPD SHARING:
Plan to Share IPD: No